CLINICAL TRIAL: NCT05865730
Title: A Phase 1/2 Study of Oncobax®-AK Administered in Combination With Immunotherapy To Patients With Advanced Solid Tumors
Brief Title: A Study of Oncobax®-AK in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EverImmune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EV-2101
Record Dates: First submitted 2023-03-20; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: 1 cohort of patients with NSCLC recruited in parallel to 1 cohort recruiting RCC patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 2 - NSCLC (Experimental): Oncobax-AK (1 capsule) will be administered daily until PD< excessive toxicity or withdrawal of consent
  Interventions: Other: Live Bacterial Product - Akkermansia muciniphila
- Phase 2 -RCC (Experimental): Oncobax-AK (1 capsule) will be administered daily until PD< excessive toxicity or withdrawal of consent
  Interventions: Other: Live Bacterial Product - Akkermansia muciniphila

INTERVENTIONS:
Other: Live Bacterial Product - Akkermansia muciniphila — Oral administration of Oncobax-AK to patients deficient in Akkermansia by stool metagenomic analysis.

SUMMARY:
Akkermansia muciniphila is a naturally occurring bacterium found in the healthy human gastrointestinal tract.

Analysis of the gut microbiota of NSCLC or RCC patients shows that the presence of Akkermansia is associated with the clinical efficacy of immunotherapy. In preclinical models, oral administration of the Akkermansia p2261 strain reverses resistance to PD-1 blockade. In the clinical setting, it is therefore hypothesized that the oral administration of Oncobax®-AK to cancer patients under immunotherapy, but whose gut microbiota is deficient in Akkermansia will restore / improve the efficacy of immunotherapy in patients with NSCLC or RCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Histologically confirmed Stage IV non-squamous NSCLC or clear cell RCC
3. NSCLC-specific criterion: Best tumor response (by iRECIST) as Stable Disease
4. NSCLC-specific criterion: PD-L1 expression > 50%
5. ECOG Performance Status = 0-1
6. Negative stool PCR test for Akkermansia
7. At least one measurable lesion per iRECIST
8. Hemoglobin ≥ 100 g/L
9. Albumin > 35 g/L
10. Signed informed consent

Exclusion Criteria:

1. Symptomatic brain metastases
2. AST or ALT > 5 x ULN
3. Calculated creatinine clearance < 45 ml/min
4. Auto-immune diseases requiring systemic therapy
5. Immunosuppressive therapy (> 10 mg prednisone/day equivalent)
6. Radiotherapy (> 30 Gy) to the lung(s) within 6 months of signed informed consent
7. Active infection
8. Co-morbidities that may increase the risk of treatment-related adverse events
9. Pregnancy
10. Inability to comply with protocol-specific assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 9 months
  iRECIST

SECONDARY OUTCOMES:
Progression-free survival | 9 months
  iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Barlesi, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (4):
- CHU Ambroise Paré, Mons, Belgium
- France (3):
  - Centre Georges Francois Leclerc, Dijon
  - Institut Gustave Roussy, Paris
  - ICANS - Institut de cancérologie Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derosa L, Routy B, Thomas AM, Iebba V, Zalcman G, Friard S, Mazieres J, Audigier-Valette C, Moro-Sibilot D, Goldwasser F, Silva CAC, Terrisse S, Bonvalet M, Scherpereel A, Pegliasco H, Richard C, Ghiringhelli F, Elkrief A, Desilets A, Blanc-Durand F, Cumbo F, Blanco A, Boidot R, Chevrier S, Daillere R, Kroemer G, Alla L, Pons N, Le Chatelier E, Galleron N, Roume H, Dubuisson A, Bouchard N, Messaoudene M, Drubay D, Deutsch E, Barlesi F, Planchard D, Segata N, Martinez S, Zitvogel L, Soria JC, Besse B. Intestinal Akkermansia muciniphila predicts clinical response to PD-1 blockade in patients with advanced non-small-cell lung cancer. Nat Med. 2022 Feb;28(2):315-324. doi: 10.1038/s41591-021-01655-5. Epub 2022 Feb 3. PMID 35115705
- [Background] Derosa L, Routy B, Fidelle M, Iebba V, Alla L, Pasolli E, Segata N, Desnoyer A, Pietrantonio F, Ferrere G, Fahrner JE, Le Chatellier E, Pons N, Galleron N, Roume H, Duong CPM, Mondragon L, Iribarren K, Bonvalet M, Terrisse S, Rauber C, Goubet AG, Daillere R, Lemaitre F, Reni A, Casu B, Alou MT, Alves Costa Silva C, Raoult D, Fizazi K, Escudier B, Kroemer G, Albiges L, Zitvogel L. Gut Bacteria Composition Drives Primary Resistance to Cancer Immunotherapy in Renal Cell Carcinoma Patients. Eur Urol. 2020 Aug;78(2):195-206. doi: 10.1016/j.eururo.2020.04.044. Epub 2020 May 4. PMID 32376136